CLINICAL TRIAL: NCT01125423
Title: An Open-Label Pilot Study to Assess Potential Mechanisms for Fibromyalgia in Peripheral Tissue Innervation That Could Predict Therapeutic Responsiveness to Milnacipran
Brief Title: Study of Fibromyalgia Treated With Milnacipran
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albany Medical College (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Charles Argoff, Principal Investigator, Albany Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIL2009-FFMS
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Fibromyalgia
Keywords: Female; age 18 to 70
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects with Fibromyalgia (Active Comparator): Subjects with Fibromyalgia have skin biopsies taken from the dominant trapezius and palm. Subjects will receive an eight week supply of milnacipran to be titrated 12.5 mg x one day, 12.5 mg twice a day x 2 days, 25mg twice daily for 4 days, then 50mg twice a day x 7 weeks.
  Interventions: Drug: Milnacipran; Procedure: Skin biopsy
- Control subjects without Fibromyalgia (Other): Subjects without Fibromyalgia have skin biopsies taken from the dominant trapezius and palm.
  Interventions: Procedure: Skin biopsy

INTERVENTIONS:
Drug: Milnacipran — Subject with Fibromyalgia will then be titrated onto milnacipran over 8 days to subject reported optimal pain control or a maximal dose of 100mg/day per package insert. Subjects will be permitted to increase or decrease their dosing at any time during the study per MD discretion in order to maintain optimal pain control.
  Other Names: Savella
  Arms: Subjects with Fibromyalgia
Procedure: Skin biopsy — Subjects with Fibromyalgia will have 3 mm skin biopsies obtained from the dominant trapezius and the glabrous hypothenar area of the hand.
Procedure: Skin Biopsy — Control Subjects will have 3 mm skin biopsies obtained from the dominant trapezius and the glabrous hypothenar area of the hand.

SUMMARY:
The purpose of this study is to examine the characteristics of the nerves and the small veins in the skin of people with fibromyalgia. This information will then be used to identify possible processes in the skin that may help explain why some people feel pain relief with the study drug (milnacipran) and others do not. The investigators expect to learn more about the pathophysiology of fibromyalgia and the way in which milnacipran acts on these patients. The investigators hypotheses are:

1. The pathophysiologic basis of fibromyalgia in some patients may be due to a biochemical and/or morphological pathology among the sensory innervation.
2. Fibromyalgia patients may have different sites of innervation.
3. Milnacipran may have a therapeutic effect on some fibromyalgia patients.
4. Abnormalities in fibromyalgia patients may predict the likelihood of a good response to milnacipran.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18-70
* fulfill the ACR criteria for FMA (wide spread pain for a least 3 months and pain in at least 11 or 18 tender point sites.
* VAS score greater that 40mm at Screening and Randomization visits.

Exclusion Criteria:

* History of clinically significant liver disease, serious peripheral vascular disease, a blood clotting disorder, or any other medical condition felt to be exclusionary by the investigator.
* Allergy to lidocaine
* Unwillingness to sign informed consent or any other reasons for which the investigator feels the subject cannot complete the study
* Women who are pregnant, breastfeeding or trying to become pregnant
* Active cancer with the previous two years except treated basal cell carcinoma of the skin.
* presence of dermatological or neurological condition that could interfere with the interpretation of the skin biopsy or QST
* Co-existing conditions that can produce chronic widespread pain
* Presence of uncontrolled or severe depression
* Patients with Worker's Compensation, pending Worker's Compensation,
* any ongoing litigation or disability claims due to fibromyalgia or any other source of pain, or currently receiving monetary compensation as a result of any of the above.
* presence of uncontrolled narrow-angle glaucoma

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of milnacipran will be determined by neurological and pain assessments | 10 weeks
  Patients will be evaluated prior to being started on milnacipran and again after 8 weeks. We will use data from VAS scores, sleep diaries and quantitative sensory testing.

CONTACTS AND LOCATIONS:
Overall Officials: Charles E. Argoff, MD, Principal Investigator — Neurosciences Institute, Albany Medical College
Locations (1):
- Upstate Clinical Research, LLC, Albany, New York, United States